CLINICAL TRIAL: NCT02393833
Title: Assessment of Vascular Endothelial Growth Factor (VEGF), Soluble Her2 Protein (NRP, Neu-Related Protein), and Vascular Cellular Adhesion Molecule-1 (VCAM-1) in Serum Samples of Patients Participating in Trial IBCSG 22-00
Brief Title: IBCSG Trial 22-00 Serum Substudy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sufficient statistical power cannot be met due to low samples size
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IBCSG 22-00 Serum Substudy; 2005-005666-36 (EudraCT Number); IBCSG 22-00 (Other: IBCSG)
Record Dates: First submitted 2014-03-12; First posted 2015-03-19 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: Vascular endothelial growth factor (VEGF); Vascular cell adhesion molecule-1 (VCAM-1); HER2-ECD
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction chemotherapy (Active Comparator): Approved induction CT regimen after randomization
  Interventions: Procedure: Blood samples collection
- Induction chemotherapy followed by CM maintenance (Experimental): Approved induction chemotherapy followed by 12 months of CM maintenance
  Interventions: Procedure: Blood samples collection

INTERVENTIONS:
Procedure: Blood samples collection — Blood samples to be collected at the following time points:
  1. Baseline, (after the completion of induction chemotherapy and, if randomized to CM maintenance, before start of CM maintenance.)
  2. Months 12, 18 and 36 after start of induction chemotherapy
  3. At time of confirmatory evidence of progression

SUMMARY:
The serum protein research study is a substudy of the core study 'Maintenance Chemotherapy in Hormone Non-responsive Breast Cancer'. This substudy is an evaluation of blood proteins and their relationship to breast cancer treatment. It will assess the levels of Vascular Endothelial Growth Factor (VEGF), Soluble HER2 Protein (NRP, neu-related protein) and Vascular Cellular Adhesion Molecule-1 (VCAM-1) in serum samples of patients' blood at different time points. The goal is to evaluate differences in serum levels between patients receiving the maintenance chemotherapy and those who do not. The serum levels will be also examined to determine if they vary during the three year period of evaluation. In addition, the serum levels of patients who have a recurrence of their breast cancer will be compared with those who remain disease free. The information obtained from these studies will enable breast cancer physicians to better tailor therapies for future patients.

DETAILED DESCRIPTION:
The Serum Substudy will assess the levels of Vascular Endothelial Growth Factor (VEGF), Soluble HER2 Protein (NRP, neu-related protein) and Vascular Cellular Adhesion Molecule-1 (VCAM-1) in patients' serum samples at different time points.

VEGF: Angiogenesis plays a central role in tumor progression of solid neoplasia. The switch from the avascular to the vascular phase is generally accompanied by rapid primary tumor growth and local invasiveness. Furthermore, angiogenesis is also necessary both at the beginning and end of the development of distant metastasis and is implicated in the phenomenon of dormant micrometastases. Antiangiogenic peptides may be altered in the serum or urine of cancer patients. In a study of 144 breast cancer patients, angiogenic protein basic fibroblast growth factor was abnormally elevated in the urine in 29% of cases and in the serum in 10%. Another angiogenic protein, vascular endothelial factor (VEGF), was abnormally elevated in the serum in over 70% of these breast cancer patients (4). Since platelets bind VEGF, platelet values will also be assayed.

HER2-ECD: No data are available regarding the presence of serum HER2-ECD (NRP) levels in c-erbB2 negative tumors, but the extracellular domain of the c-erbB2 oncogene product (NRP) is detectable in sera of 30-60% of patients with cerbB2 positive tumors. Many reports have correlated the elevated serum levels of the cerbB2 with gene amplification and c-erbB2 overexpression in tumor. These data support the hypothesis that the level of NRP protein can reflect the presence of c-erbB2 positive cells and that modification of the factor can predict a decrease of c-erbB2 positive cells during standard adjuvant chemotherapy. Moreover, change in the detectable NRP during the maintenance phase can suggest a possible modification in the biology and/or behaviour of hypothetic micrometastasis.

VCAM-1: In tumors, endothelial VCAM-1 play a major role in the adhesion of leukocytes to the endothelium, suggesting a relationship between cellular adhesion and angiogenesis. Soluble VCAM-1 has been implicated in the mediation of angiogenesis and some studies support the hypothesis that VCAM-1 provides surrogate markers for endothelial activation and angiogenesis occurring during cancers. Recently, VCAM-1 serum levels have been associated with microvessel density and response to endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be randomized to the core protocol. Written informed consent for the serum substudy must be signed and dated by the patient and investigator
* Patient must not have begun CM maintenance (if randomized to CM maintenance)

Exclusion Criteria:

* Patient not randomized to the core protocol
* Patient already begun CM maintenance (if randomized to CM maintenance)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2002-06; Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 18 months in serum VEGF values | 18 months
  To evaluate differences from baseline (after completion of induction chemotherapy but before commencement of CM Maintenance for patients randomized to CM Maintenance) to 18 months after the start of induction chemotherapy in serum VEGF values between patients in the Observation Group and those in the low dose Cyclophosphamide Methotrexate (CM) Maintenance Group.
Change from baseline to 18 months in serum VCAM-1 values | 18 months
  To evaluate differences from baseline (after completion of induction chemotherapy but before commencement of CM Maintenance for patients randomized to CM Maintenance) to 18 months after the start of induction chemotherapy in serum VCAM-1 values between patients in the Observation Group and those in the low dose Cyclophosphamide Methotrexate (CM) Maintenance Group.
Change from baseline to 18 months in serum NRP values | 18 months
  To evaluate differences from baseline (after completion of induction chemotherapy but before commencement of CM Maintenance for patients randomized to CM Maintenance) to 18 months after the start of induction chemotherapy in serum NRP values between patients in the Observation Group and those in the low dose Cyclophosphamide Methotrexate (CM) Maintenance Group.

SECONDARY OUTCOMES:
Change from baseline to 12 and 36 months in serum VEGF values | 12 & 36 months
  To compare the differences from baseline to 12 and 36 months in serum VEGF values in the two randomized groups.
Change from baseline to 12 and 36 months in serum VCAM-1 values | 12 & 36 months
  To compare the differences from baseline to 12 and 36 months in serum VCAM-1 values in the two randomized groups.
Change from baseline to 12 and 36 months in serum NRP values | 12 & 36 months
  To compare the differences from baseline to 12 and 36 months in serum NRP values in the two randomized groups.
Change in serum VEGF values from last measurement before progression to measurement at time of confirmatory evidence of progression | Baseline,12-, 18- or 36-months & progression
  To compare VEGF values before and after progression in the two randomized groups.
Change in serum VCAM-1 values from last measurement before progression to measurement at time of confirmatory evidence of progression | Baseline,12-, 18- or 36-months & progression
  To compare VCAM-1 values before and after progression in the two randomized groups.
Change in serum NRP values from last measurement before progression to measurement at time of confirmatory evidence of progression | Baseline,12-, 18- or 36-months & progression
  To compare NRP values before and after progression in the two randomized groups.

CONTACTS AND LOCATIONS:
Overall Officials: Aron Goldhirsch, Prof., Study Chair — IEO Milano; Giuseppe Viale, Prof., Study Chair — IEO Milano
Locations (3):
- Istituto Europeo di Oncologia (IEO, Milan, Italy
- Ibadan, Nigeria
- Lima, Peru

REFERENCES:
- [Background] Kern FG, Lippman ME. The role of angiogenic growth factors in breast cancer progression. Cancer Metastasis Rev. 1996 Jun;15(2):213-9. doi: 10.1007/BF00437474. No abstract available. PMID 8842493
- [Background] Gasparini G. Clinical significance of the determination of angiogenesis in human breast cancer: update of the biological background and overview of the Vicenza studies. Eur J Cancer. 1996 Dec;32A(14):2485-93. doi: 10.1016/s0959-8049(96)00376-0. No abstract available. PMID 9059337
- [Background] Revillion F, Hebbar M, Bonneterre J, Peyrat JP. Plasma c-erbB2 concentrations in relation to chemotherapy in breast cancer patients. Eur J Cancer. 1996 Feb;32A(2):231-4. doi: 10.1016/0959-8049(95)00568-4. PMID 8664033
- [Background] Byrne GJ, Ghellal A, Iddon J, Blann AD, Venizelos V, Kumar S, Howell A, Bundred NJ. Serum soluble vascular cell adhesion molecule-1: role as a surrogate marker of angiogenesis. J Natl Cancer Inst. 2000 Aug 16;92(16):1329-36. doi: 10.1093/jnci/92.16.1329. PMID 10944555
- See also: Sponsor — http://www.ibcsg.org/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2005-11-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT02393833/Prot_SAP_000.pdf